CLINICAL TRIAL: NCT01960127
Title: Effects of Aerobic Training on Exercise Capacity in Patients With Advanced Cirrhosis 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LZPTMH2.0
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental): Supervised aerobic training 3 times per week for 8 weeks (30-60 minute sessions)
  Interventions: Behavioral: Aerobic Exercise
- Usual Care Group (Placebo Comparator): These patients will continue with their normal daily activity ad will not be provided with supervised aerobic exercise training during the study period.
  Interventions: Behavioral: No Intervention

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise
  Arms: Aerobic Exercise
Behavioral: No Intervention — No Intervention
  Arms: Usual Care Group

SUMMARY:
Cirrhosis is associated with a reduction in muscle mass and exercise capacity. This has an impact on morbidity and mortality. Regular aerobic exercise training is a proven effective therapy to improve exercise capacity in healthy and clinical populations. The effect of this training has not yet been evaluated in the decompensated cirrhosis patient population. The safety of this intervention also requires further study. Using a randomized controlled design, the investigators aim to determine the safety and efficacy of eight weeks of aerobic exercise training on aerobic capacity, functional performance, and muscle mass in decompensated cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and ≤ 70 years
* Cirrhosis
* Child Pugh class B or C
* If required, primary or secondary variceal prophylaxis in place

Exclusion Criteria:

* Post-liver transplantation
* Hepatocelluar carcinoma beyond transplant criteria
* Active non-hepatocelluar carcinoma malignancy
* Significant cardiac disease
* Hemoglobin (<80 g/L)
* Oxygen saturation at rest <95%
* Known myopathy
* Chronic renal failure on dialysis
* Physical impairment making it impossible to ride an exercise bike or treadmill
* Orthopedic abnormality preventing exercise training
* HIV infection
* Patient unwilling to consent to study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change in peak exercise pulmonary oxygen uptake (peak V02) | Baseline (day1) and Study End (8 weeks)

SECONDARY OUTCOMES:
Change in muscle mass as measured by thigh ultrasound | Baseline (day 1) and Study End (8 weeks)
Change in quality of life-Chronic Liver Disease Questionnaire | Baseline (day1) and Study End (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haykowsky, PhD, Study Director — University of Alberta
Locations (1):
- University of Alberta, Mazankowski Heart Institute, Edmonton, Alberta, Canada